CLINICAL TRIAL: NCT03374566
Title: Screening for Immunodeficiency Diseases in Patients With Severe Epstein-Barr Virus Infection
Brief Title: Immunodeficiency for Severe Epstein-Barr Virus Infection
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jinqiao Sun, Professor, Children's Hospital of Fudan University
Other Study IDs: EBV
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Epstein-Barr Virus Infections; Immunodeficiency
Keywords: Epstein-Barr Virus Infections; Immunodeficiency; Screening; Immunologic Function
MeSH Terms: conditions — Epstein-Barr Virus Infections; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Heparinized peripheral blood is obtained from patients with severe EBV infections. Samples is performed after parents' information and consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screened patients: Immunodeficiency screening: Heparinized peripheral blood is obtained from patients with severe EBV infections for immunological function assays and genetic analysis, when current screening is performed after parents' information and consent.

SUMMARY:
The purpose of this study is to investigate the immune responses associated with Epstein-Barr virus infections, and to find out the possible immunodeficiency that may be linked to severe Epstein-Barr virus infections.

DETAILED DESCRIPTION:
Epstein-Barr virus (EBV) belongs to herpesviridae family, which infects more than 90% of the population. EBV infection is usually asymptomatic and establishes lifelong persistence in the host, although primary infection later than adolescence frequently results in infectious mononucleosis (IM). Rarely, individuals may develop a subgroup of EBV-associated life threatening complications (including liver dysfunction, haemophagocytosis and malignancy).

Although EBV-infected B cells have the potential for proliferation, they are effectively removed by the EBV-specific cytotoxic T cells (CTL). In the immunocompetent hosts, natural killer (NK) cells and antigen-specific cluster designation 8 (CD8+) T-cells play an important role in inhibiting progression of primary EBV infection by granule-mediated cytotoxicity. The immune system is necessary to control the virus-induced transformation and the B-cell unlimited proliferation.

Primary immunodeficiency are a heterogeneous group of hereditary diseases that are associated with compromised immune responses. There are a number of immunodeficiency resulting in inability of immune system to control EBV infection, for example X-linked Lymphoproliferative disease (XLP)/signaling lymphocyte activation molecule (SLAM)-associated protein (SAP) deficiency, X-linked inhibitor of apoptosis (XIAP) deficiency, cluster of differentiation antigen 27 (CD27) deficiency, interleukin-2-inducible T-cell kinase (ITK) deficiency, and so on. Whereas, some other clinical states associated with EBV-susceptibility remain largely unknown. Rare EBV-infected individuals without apparent immunodeficiency also present with persistent IM-like symptoms, hepatosplenomegaly, liver dysfunction, lymphadenopathy and haemophagocytic lymphohistiocytosis.

Patients presenting with severe EBV infections should be focused on early identification of a possible primary immunodeficiency or a chronic active EBV infection clinical condition (CAEBV) and haemophagocytic lymphohistiocytosis(HLH). Immunological phenotyping of NK-, T- and B-cell differentiation, and functional assays including cytotoxic cell killing function and cytotoxic granule release, provide a useful identification for clinical conditions inability to control EBV infections. Genomic DNA is isolated from peripheral blood mononuclear cells and will be amplified to screen for possible immunodeficiency.

The reasons for those patients inability to control the EBV infection are still unknown. However no effective treatment is currently available, those patients might benefit from early hematopoietic stem cell transplantation (HSCT). Through this study, we hope to identify the unknown immune immunodeficiency and pathophysiology of those EBV-associated conditions. The investigators propose to help make early diagnosis and develop effective therapies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age：birth to 18 years 2. Severe Epstein-Barr Virus infection

Exclusion Criteria:

* 1. Lack of parental consent

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We will evaluate immunodeficiency incidence in patients with severe EBV infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Immunodeficiency incidence in patients with severe EBV infection | 5 years
  We will investigate immunodeficiency incidence in patients with severe EBV infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jinqiao Sun, Ph.D.,M.D, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Worth AJ, Houldcroft CJ, Booth C. Severe Epstein-Barr virus infection in primary immunodeficiency and the normal host. Br J Haematol. 2016 Nov;175(4):559-576. doi: 10.1111/bjh.14339. Epub 2016 Oct 17. PMID 27748521
- [Background] Shabani M, Nichols KE, Rezaei N. Primary immunodeficiencies associated with EBV-Induced lymphoproliferative disorders. Crit Rev Oncol Hematol. 2016 Dec;108:109-127. doi: 10.1016/j.critrevonc.2016.10.014. Epub 2016 Nov 2. PMID 27931829
- [Background] Palendira U, Rickinson AB. Primary immunodeficiencies and the control of Epstein-Barr virus infection. Ann N Y Acad Sci. 2015 Nov;1356:22-44. doi: 10.1111/nyas.12937. Epub 2015 Sep 28. PMID 26415106
- [Background] Taylor GS, Long HM, Brooks JM, Rickinson AB, Hislop AD. The immunology of Epstein-Barr virus-induced disease. Annu Rev Immunol. 2015;33:787-821. doi: 10.1146/annurev-immunol-032414-112326. Epub 2015 Feb 11. PMID 25706097
- [Background] Fujiwara S, Kimura H, Imadome K, Arai A, Kodama E, Morio T, Shimizu N, Wakiguchi H. Current research on chronic active Epstein-Barr virus infection in Japan. Pediatr Int. 2014 Apr;56(2):159-66. doi: 10.1111/ped.12314. PMID 24528553
- [Background] Eligio P, Delia R, Valeria G. EBV Chronic Infections. Mediterr J Hematol Infect Dis. 2010 Aug 10;2(1):e2010022. doi: 10.4084/MJHID.2010.022. PMID 21415952